CLINICAL TRIAL: NCT00908284
Title: Atherosclerotic Risk and Response to Exercise Intervention in HIV+ Children
Brief Title: Evaluating an Exercise Program to Reduce Cardiovascular Risk Factors in Children Infected With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Tracie L. Miller, MD, Professor of Pediatrics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20030814; 1R01HL095127-01 (NIH)
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: HIV; Acquired Immunodeficiency Syndrome; Cardiovascular Diseases
Keywords: AIDS; Acquired Immune Deficiency Syndrome Virus; Human Immunodeficiency Virus; Exercise Physiology; Endothelial Dysfunction
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiovascular Diseases | interventions — Resistance Training; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Participants will take part in a 12-week control group.
  Interventions: Behavioral: Control Group
- Exercise Program (Experimental): Participants will take part in a 12-week exercise program.
  Interventions: Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Exercise Program — Participants will exercise in the study exercise laboratory for 1 hour on 2 nonconsecutive days a week for 12 weeks. The program will consist of a warm-up with flexibility exercises, aerobic conditioning, a muscular circuit, and a cool-down period with flexibility training.
  Arms: Exercise Program
Behavioral: Control Group — Participants will attend group sessions once a week for 12 weeks to watch videos, including some exercise videos, and play games that do not require physical activity.
  Arms: Control Group

SUMMARY:
People infected with HIV are now living longer lives because of the use of highly active antiretroviral therapy (HAART). However, HAART medications have been shown to increase the risk of cardiovascular disease and metabolic dysfunction in adults. More research is needed on the effect of HAART in children. The purpose of this study is to assess cardiovascular risk factors in children infected with HIV who receive HAART medications and to determine the effectiveness of an exercise program on cardiovascular outcomes in these children.

DETAILED DESCRIPTION:
People infected with HIV are now living longer and healthier lives than HIV-infected people of previous generations because of the widespread use of HAART medications. However, as HIV infection becomes a more chronic illness, rather than a fatal disease, researchers are beginning to identify the long-term complications of HIV infection and its treatment. Adults infected with HIV are increasingly developing the following: hyperlipidemia and dyslipidemia, both of which are associated with high cholesterol levels; endothelial dysfunction; insulin resistance; and changes in body composition, including increased obesity levels and an increase in central body fat. These conditions are all associated with an increased risk of cardiovascular disease. More research is needed to examine how children infected with HIV who are receiving HAART may be affected by these conditions. In this study, researchers will examine children infected with HIV who are receiving HAART (as well as a control group of children who are not infected with HIV) to evaluate vascular function and inflammation over time and how they affect body composition, fat redistribution, insulin resistance, hyperlipidemia, growth, nutrition, bone metabolism, and disease severity. This study will also evaluate the effectiveness of an exercise program on vascular function and cardiovascular outcomes in children infected with HIV who are receiving HAART.

There are two parts to this study. In Part 1, children infected with HIV and their siblings and friends who are not infected with HIV will attend study visits every 6 months for 3 years. At select visits, the following study procedures will occur: medical history review; physical exam; blood collection; body measurements; questionnaires regarding diet, quality of life, and activity levels; and an echocardiogram to obtain images of the heart.

In Part 2 of the study, a portion of participants from Part 1 of the study who are infected with HIV will be randomly assigned to take part in a 12-week exercise program or a control group. At a baseline study visit, all participants will undergo a medical history review, fitness testing, body measurements, muscle and fat measurements, blood collection, echocardiogram, questionnaires to assess quality of life and activity levels, and an ultrasound of the brachial artery (on the upper arm) and carotid artery (on the neck) to measure artery size.

Participants in the exercise program will exercise (e.g., walking, running, cycling, stretching, and weight training) for 1 hour at the study exercise laboratory 2 days a week for 12 weeks. If participants cannot come to the laboratory, they may exercise at home, under the guidance of study researchers. Participants will wear a pedometer on select days and keep an activity log to record how far they walk. At the end of the 12-week program, participants will undergo repeat baseline testing. They will also receive a written, personalized exercise program that they can follow on their own. Participants will receive weekly phone calls from study researchers and will attend study visits once a month for 3 months for follow-up and monitoring. Baseline testing will occur again at the end of the 3-month follow-up period.

Participants in the control group will attend group sessions once a week for 12 weeks at which time they will watch videos, including some exercise videos, and play games that do not require physical activity. At the end of Week 12, participants will undergo repeat baseline testing. They will then have the option of taking part in the exercise program.

ELIGIBILITY:
Inclusion Criteria for Part 1 of the Study:

HIV-Infected Children:

* Must be between 2 weeks and 25 years old with known perinatally acquired HIV infection
* Stable medical regimen for at least 3 months before study entry
* Has not used antihypertensive, hypoglycemic, or lipid-lowering medications
* Active opportunistic infection in the 3 months before study entry
* Willing to participate in the study and sign the informed consent document

Non-HIV-Infected Siblings/Friends/General Pediatric Control Group:

* Demographically similar to HIV-infected participants
* Not known to be HIV-infected
* Meets all other entry criteria for HIV-infected participants

Exclusion Criteria for Part 1 of the Study:

* Documented diabetes mellitus managed with medications
* Heart, kidney, liver, or muscle disease
* Intercurrent illness at the time of study entry and baseline testing (person can be enrolled when the illness is resolved [e.g., upper respiratory infection])

Inclusion Criteria for Part 2 of the Study:

* Must be enrolled in Part 1 of the study
* Must be between 6 and 25 years old
* Willing to participate in the exercise program and sign the informed consent document
* Has medical clearance from physician to participate in the study

Exclusion Criteria for Part 2 of the Study:

* Unable to perform or understand exercise program
* Currently taking medications that would prohibit participation in exercise programs (e.g., coumadin, heparin)
* Heart, kidney, liver, or muscle disease
* Anabolic steroid use in the 3 months before study entry (e.g., growth hormone)
* Malignant arrhythmia
* Has a pacemaker
* Orthopedic problems that would prevent performance of any of the prescribed activities
* Changes in metabolic stress testing that would make the exercise program unsafe, as determined by the reporting cardiologist (i.e., ischemic changes)

Ages: 2 Weeks to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2008-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
E-selectin, vascular cell adhesion molecule-1 (VCAM-1), P-selectin, fibrinogen, plasminogen activator inhibitor-1 (PAI-1), and monocyte chemoattractant protein-1 (MCP-1) | Measured at Year 3
High sensitivity C-reactive protein (hs-CRP), interleukin-6 (IL-6), adiponectin, leptin, mitochondrial DNA (mtDNA), echocardiography, flow-mediated dilation (FMD), and carotid intima-media thickness (cIMT) | Measured at Year 3
Body mass index (BMI), dual energy x-ray absorptiometry (DXA), bioelectrical impedance analysis (BIA), resting energy expenditure (REE), bone mineral density (BMD), lipid profiles, insulin and glucose strength, and fitness measures | Measured at Year 3

SECONDARY OUTCOMES:
Age, sex, HIV disease stage, CD4 counts, viral load, and type and length of antiretroviral therapies | Measured at Year 3

CONTACTS AND LOCATIONS:
Overall Officials: Tracie L. Miller, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Department of Pediatrics, Division of Clinical Research, Batchelor Children's Research Institute, Miami, Florida, United States